CLINICAL TRIAL: NCT06832306
Title: A Clinical Study Evaluating Temporary Transvenous Diaphragm Neurostimulation in Mechanically Ventilated Patients With Acute Hypoxemic Respiratory Failure
Brief Title: STimulation to Activate RespIration
Acronym: STARI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lungpacer Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-600; 75A0123C00021 (Other Grant/Funding Number: Biomedical Advanced Research and Development Authority (BARDA))
Record Dates: First submitted 2025-02-06; First posted 2025-02-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-05

CONDITIONS: ARDS (Moderate or Severe); AHRF; Mechanically Ventilated ICU Patients
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: 2:1 Randomization treatment to control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment (Experimental): Treatment group subjects will have the Catheter placed percutaneously into the left jugular vein or left subclavian vein. Mapping will identify the electrodes that stimulate the phrenic nerves and enable diaphragm contraction using the AeroNova Console. The stimulation level will be titrated to target a level of diaphragm activation equivalent to resting quiet breathing by adjusting the stimulation frequency and amplitude. Subjects will receive continuous stimulation plus standard of care lung-protective ventilation.
  Interventions: Device: Phrenic Nerve Stimulation
- Control (No Intervention): Standard of Care - Lung-protective ventilation

INTERVENTIONS:
Device: Phrenic Nerve Stimulation — During controlled MV when patients are not breathing, continuous diaphragm neurostimulation-assisted ventilation (DNAV) will be delivered in synchrony with each ventilator-delivered breath.
  Other Names: Diaphragm neurostimulation-assisted ventilation (DNAV)
  Arms: Treatment

SUMMARY:
Multi-center, randomized, controlled, open-label Phase 2 feasibility trial. Subjects on mechanical ventilation (MV) for acute hypoxemic respiratory failure (AHRF) with lung injury (including subjects who meet criteria for acute respiratory distress syndrome (ARDS)) will be randomized 2:1 to diaphragm neurostimulation-assisted ventilation (DNAV) using the AeroNova System plus lung-protective ventilation (Treatment) vs. lung-protective ventilation alone (Control).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years or older, and
2. Able to provide informed consent or have a legally authorized representative (LAR) / Substitute Decision Maker (SDM) who can provide consent, and
3. Have acute onset of new respiratory symptoms or dysfunction within the 2 weeks before onset of need for respiratory support, and
4. Have arterial hypoxemia defined by one of:

   * PaO2:FiO2 ratio ≤300 mm Hg on PEEP ≥5 cm H2O, or
   * In the absence of an available arterial blood gas, SpO2 ≤97% on FiO2 ≥0.5 and PEEP ≥5 cm H2O with reliable SpO2 trace for the 2 hours immediately preceding eligibility assessment (this correlates to an upper limit of SpO2:FiO2 ratio of 316%) or
   * Are receiving pulmonary vasodilators for acute hypoxemia, or
   * Are being ventilated in the prone position for acute hypoxemia, and
5. Have been mechanically ventilated for AHRF in the ICU for <96 hours at the time of enrolment, and
6. Are expected to require invasive mechanical ventilation ≥48 hours after enrollment in the opinion of the treating clinician

Exclusion Criteria:

1. Hypoxemia is primarily attributable to acute exacerbation of chronic obstructive pulmonary disease, status asthmaticus, cardiogenic pulmonary edema, or pulmonary embolism.
2. Underlying chronic parenchymal lung disease that may make recovery/extubation a challenge (e.g., COPD, pulmonary fibrosis).
3. Broncho-pleural fistula at the time of eligibility assessment.
4. Require extracorporeal membrane oxygenation.
5. Pre-existing neurological, neuromuscular or muscular disorder or known phrenic nerve injury that could affect the respiratory muscles.
6. BMI >70 kg/m2.
7. Contraindications to left internal jugular vein or left subclavian vein catheterization (e.g., infection at the access site, known central venous stenosis, septic thrombophlebitis, left internal jugular ECMO cannula in situ, poor target vessels).
8. Patient expected to transition to fully palliative care within 72 hours of enrollment.
9. Chronic severe liver disease (e.g., Child-Pugh Score ≥10)
10. Treating clinician deems enrollment not clinically appropriate.
11. Currently enrolled in any other study of an investigational drug or device, which may affect the outcomes of the current study.
12. Any electrical device (implanted or external) that may be prone to interaction with or interference from the AeroNova System, including neurological pacing/stimulator devices and cardiac pacemakers and defibrillators.
13. Known or suspected to be pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Successful device insertion, mapping, and initiation of stimulation within 18 hours of meeting readiness-to-stimulate criteria | Within 18 hours of meeting readiness to stimulate criteria
Stimulation delivered on >50% of ventilator-triggered breaths (ascertained from continuous recordings stored in the Console) | 30 days
Rehabilitation sessions delivered at least once per day on >50% of days when the patient was breathing in assisted (patient-triggered) mechanical ventilation | 30 days

SECONDARY OUTCOMES:
Unanticipated serious adverse device events (USADE) and incidence of device- or procedure-related SAEs in the Treatment group | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ewan Goligher, MD, PhD, FRCPC, Principal Investigator — Toronto General Hospital
Locations (6):
- United States (5):
  - University of California San Diego, La Jolla, California
  - Louisiana State University Health Sciences, Shreveport, Louisiana
  - Cleveland Clinic, Cleveland, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - Prisma Health, Columbia, South Carolina
- University Health Network (UHN), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes